CLINICAL TRIAL: NCT00002604
Title: Phase I Trial of O6 Benzylguanine and BCNU; A Biochemical Modulation Trial Based Upon Depletion of O6 Alkylguanine DNA Alkyltransferase Directed DNA Repair
Brief Title: O(6)-Benzylguanine and Carmustine in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James K.V. Willson, Jr. MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1994; U01CA062502 (NIH); CWRU-ICC-1994; NCI-T94-0022D
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — O(6)-benzylguanine; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: O6-benzylguanine — Patients receive BG IV over 1 hour during week 1, and then BG IV over 1 hour during week 3. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
Drug: carmustine — After one hour of receiving BG patients receive BCNU IV over 1 hour during week 3. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Other Names: BCNU
Drug: chemosensitization/potentiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of O(6)-benzylguanine and carmustine in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the biochemical modulation dose l of O6-benzylguanine (BG), defined as the dose at which baseline O6-alkylguanine DNA alkyltransferase (AGT) activity in circulating peripheral blood mononuclear cells (PBMC) decreases by greater than 90% in patients with advanced solid tumors at 2 hours after BG infusion. II. Determine the biochemical modulation dose t/18 (BMDt/18) of BG, defined as the dose at which AGT activity in human metastatic tumor tissue decreases to undetectable levels at 18 hours after BG infusion. III. Determine the maximum tolerated dose of carmustine (BCNU) when administered with BG at the BMDt/18 in these patients. IV. Determine the toxicities of BG and BCNU in these patients. V. Determine the pharmacokinetic parameters of BG administered at the BMDt/18, and determine any effects of BCNU on BG pharmacokinetics. VI. Assess any antitumor response in patients with metastatic solid tumors treated with this regimen. VII. Determine the effect of lower, more frequent bolus doses or a continuous infusion of BG on the depletion of AGT activity in PBMC and tumor tissue in these patients. VIII. Determine the pharmacokinetics of BG in lower, more frequent bolus doses or continuous infusion.

OUTLINE: This is a dose escalation study of 06-benzylguanine (BG) and carmustine (BCNU). Patients receive BG IV over 1 hour during week 1, and then BG IV over 1 hour followed 1 hour later by BCNU IV over 1 hour during week 3. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 1-3 patients receive escalating doses of BG until the biochemical modulation dose l (BMDl) is determined. The BMDl is defined as the dose at which baseline O6-alkylguanine DNA alkyltransferase (AGT) activity in circulating peripheral blood mononuclear cells decreases by greater than 90% at 2 hours after BG infusion. Cohorts of 3 patients receive escalating doses of BG beginning at the BMDl until the biochemical modulation dose t/2 (BMDt/2) is determined. The BMDt/2 is defined as the dose at which AGT activity in human metastatic tumor tissue decreases by greater than 90% at 2 hours after BG infusion. Cohorts of 3 patients receive escalating doses of BG beginning at the BMDt/2 until the biochemical modulation dose t/18 (BMDt/18) is determined. The BMDt/18 is defined as the dose at which AGT activity in human metastatic tumor tissue decreases to undetectable levels at 18 hours after BG infusion. Patients then receive BG IV over 1 hour followed 1 hour later by BCNU IV over 1 hour during week 1. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of BCNU combined with BG at the BMDt/18 until the maximum tolerated dose (MTD) of BCNU is determined. The MTD of BCNU is defined as the dose preceding that at which 2 or more of 6 patients experience dose limiting toxicity. A cohort of 3 patients receives BG IV over 2 minutes and another cohort of 3 patients receives BG IV over 24 hours. An additional cohort of 6 patients receives BG IV over 24 hours and BCNU IV over 1 hour beginning 2 hours into BG infusion during week 3.

PROJECTED ACCRUAL: A total of 51 patients will be accrued for this study over 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumor for which no standard treatment exists (including surgery, radiotherapy, or systemic agents) No primary CNS malignancy No CNS metastases Only disease that can be sequentially biopsied is eligible for determination of the biochemical modulating dose that decreases AGT in tumor tissue

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Hematopoietic: WBC greater than 4,000/mm3 Absolute neutrophil count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 3 times normal Prothrombin time less than upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Calcium normal Electrolytes normal Other: Diabetes controlled by diet or insulin allowed Not pregnant Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since chemotherapy (6 weeks since mitomycin) and recovered No prior nitrosoureas Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1996-01; Primary Completion 2000-07 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
dose escalation study of 06-benzylguanine (BG) and carmustine (BCNU) | Courses (each course is 3 weeks) repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 1-3 patients receive escalating doses of BG until the biochemical modulation dose l (BMDl) is determined.

CONTACTS AND LOCATIONS:
Overall Officials: James KV Willson, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio